CLINICAL TRIAL: NCT06939881
Title: "11 For Health" in Türkiye - Effects on Physical Performance and Executive Function in 10-11-Years-Old Schoolchildren
Brief Title: "11 For Health" in Türkiye; Effect on Physical Performance and Executive Function in 10-11-Year-Olds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Namik Kemal University (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, umut canlı, Professor, Namik Kemal University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NamikemalUU
Record Dates: First submitted 2025-04-11; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Physical Activity; Executive Function (Cognition); Physical Performance
Keywords: 11 for Health in Türkiye; executive function; schoolchildren
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The study sample was determined and divided into groups using the convenience sampling method. This non-random sampling approach involves selecting participants based on the researcher's judgment, allowing for practical, fast, and cost-effective data collection. At this stage, two 5th-grade classes from the same school that met the inclusion criteria and agreed to participate were selected. One class was assigned as the control group (CG; n=29) and the other as the training group (TG; n=27).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "11 for Health" program (Experimental): "11 for Health" program training group
  Interventions: Other: "11 for Health" training group
- control group (No Intervention): Control Group; The control group continued with their regular school curriculum, which included two 45-minute physical education classes per week, and did not receive any additional intervention.

INTERVENTIONS:
Other: "11 for Health" training group — The "11 for Health" intervention consisted of two 45-minute sessions per week for 11 weeks, implemented during school hours. Each week included one session focused on football-related physical activities (e.g., passing, dribbling, shooting) and another on health education topics (e.g., hygiene, nutrition, mental well-being), both delivered in an engaging and inclusive format. The program emphasized social interaction, autonomy-supportive teaching, and real-life applicability through take-home tasks.
  Arms: "11 for Health" program

SUMMARY:
The goal of this study was to evaluate whether the school-based "11 for Health" program could improve physical performance and executive function among 10-11-year-old Turkish schoolchildren. The main questions it aimed to answer were:

Does the program enhance physical performance, including agility, balance, and vertical jump? Does it improve executive function skills such as response inhibition, problem solving, and working memory? Researchers compared students who participated in the 11-week "11 for Health" intervention to those who continued their regular school curriculum.

Participants:

A total of 56 children (28 girls and 28 boys) from 5th grade participated. The training group attended two 45-minute "11 for Health" sessions per week for 11 weeks.

Both groups were assessed before and after the intervention on physical performance (e.g., balance, agility, countermovement jump) and executive function (Go/No-Go, Tower of Hanoi, and Corsi Block tests).

DETAILED DESCRIPTION:
This study examined the impact of the school-based "11 for Health" program on the physical performance and executive function of 10-11-year-old Turkish schoolchildren. The program, developed by FIFA in collaboration with global health experts, integrates football-based physical activities with health education content. Given the growing concern over insufficient physical activity levels among children in Türkiye, the intervention sought to explore how structured school-based programs could enhance not only physical performance but also higher-order cognitive processes.

The rationale for the study stems from evidence indicating that physical activity is not only essential for maintaining cardiovascular and musculoskeletal health but also closely linked to cognitive functions such as attention, response inhibition, and planning. Executive functions are critical during late childhood as they influence academic performance, behavior regulation, and social competence.

The "11 for Health" intervention consisted of two 45-minute sessions per week for 11 weeks, implemented during school hours. Each week included one session focused on football-related physical activities (e.g., passing, dribbling, shooting) and another on health education topics (e.g., hygiene, nutrition, mental well-being), both delivered in an engaging and inclusive format. The program emphasized social interaction, autonomy-supportive teaching, and real-life applicability through take-home tasks.

Participants were divided into a training group and a control group using convenience sampling. The training group received the intervention, while the control group continued their standard physical education curriculum. Pre- and post-intervention assessments were conducted over separate days to measure changes in physical and cognitive outcomes.

Physical performance was assessed using standardized protocols to evaluate balance (static, proprioceptive, dynamic), agility (pro-agility shuttle test), and vertical jump (countermovement jump). Executive function was measured using three computer-based tasks: the Go/No-Go test (response inhibition), the Tower of Hanoi (planning/problem-solving), and the Corsi Block Test (visuospatial working memory).

The study contributes to the growing literature on school-based physical activity interventions and their multifaceted impact on children's development, offering insights relevant to both educators and policymakers seeking to optimize school curricula for health and cognitive outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Typically developing children
* Aged between 10 and 11 years
* Enrolled in the 5th grade of primary school
* Not currently taking any medication
* Provided informed consent from both the child and their parent/guardian

Exclusion Criteria:

* Having any diagnosed cardiovascular, neurological, orthopedic, or psychiatric condition
* Taking regular medication
* Outside the age range of 10-11 years
* Presence of any developmental disorder or learning disability

Ages: 10 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-06-14 (Actual)

PRIMARY OUTCOMES:
Changes in Static Balance Performance (% Score) | before and at the end of the 11-week intervention.
  Static balance was measured using the Sensbalance MiniBoard device. Participants were asked to stand still on the platform for approximately 30 seconds. The device calculated the participant's ability to maintain posture without significant sway.
Changes in Dynamic Balance Performance - Left-Right and Front-Back (% Score) | before and at the end of the 11-week intervention.
  Dynamic balance was evaluated using the Sensbalance MiniBoard through controlled weight shifting in mediolateral and anteroposterior directions.
Changes in Proprioceptive Balance Performance (% Score) | before and at the end of the 11-week intervention.
  Proprioceptive balance was assessed via subtle postural adjustments on the Sensbalance MiniBoard. Scores were automatically generated based on sway control.
Changes in Countermovement Jump Performance (cm) | before and at the end of the 11-week intervention.
  Vertical jump height was measured using an accelerometer-based system (IVMES, Ankara, Turkey) during countermovement jump (CMJ) trials. Unit of Measurement: Centimeter (cm) - Highest jump height
Changes in Agility (seconds) | before and at the end of the 11-week intervention.
  Assessed via the Pro-Agility Test (20-yard shuttle run) using photocell timing gates. The total time to complete the right-left-center shuttle sequence was recorded. Unit of Measurement: Seconds (s) - Time to complete the test
Changes in Inhibitory Control (Number of correct responses and Reaction Time (ms)) | before and at the end of the 11-week intervention.
  Inhibitory control was assessed using a computer-based Go/No-Go task, which measured participants' ability to suppress automatic motor responses. The task included 200 trials: 100 Go (letter X) and 100 No-Go (letter O) stimuli. Participants were instructed to press a button as quickly as possible for Go stimuli and withhold responses for No-Go stimuli. Key outcome variables included:
  Accuracy of correct responses to Go stimuli (AC-Go) Accuracy of correct inhibitions to No-Go stimuli (AC-NoGo) Mean reaction time for correct Go responses (Go RT)
  Unit of Measurement: Number of correct responses and reaction time in milliseconds (ms)
Changes in Planning and Problem-Solving Skills (Number of moves and seconds) | before and at the end of the 11-week intervention.
  Description: Executive function was assessed using a computer-based Tower of Hanoi task, designed to evaluate planning, problem-solving, and rule-based learning. Participants moved three disks across three pegs while following predefined rules to match a target configuration. Four outcome variables were recorded:
  Total number of moves Total time to solution (seconds) Average time per move (seconds) Latency to first move (planning time in seconds)
  Unit of Measurement: Number of moves and seconds (s)
Changes in Visuospatial Working Memory (correctly repeated number score) | before and at the end of the 11-week intervention.
  Description: The Corsi Block Test was used to evaluate visual working memory and attention. In this computerized task, participants were asked to reproduce increasingly complex sequences of illuminated blocks. The task terminated when the participant failed to correctly repeat sequences of a given length twice in a row.
  Unit of Measurement: Span score (maximum sequence length correctly repeated)

CONTACTS AND LOCATIONS:
Locations (1):
- Tekirdag Namik Kemal University, Sports Sciences Research and Development Centre, Tekirdag, Suleymanpasa 59030, Tekirdağ, Suleymanpasa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Measurements: Data obtained from physical fitness parameters (e.g., static, dynamic and proprioceptive balance, agility, countermovement jump) and executive function assessments (e.g., Go/No-Go, Tower of Hanoi, and Corsi Block tests) will be shared.
  Data Anonymization: All shared data will be fully anonymized to ensure participant confidentiality. Personal identifiers such as names, birth dates, and school affiliations will be removed. Data will be reviewed and aggregated where necessary to prevent the possibility of participant re-identification.
  Data Format: The data will be provided in standardized file formats such as CSV or Excel (.xlsx) to support compatibility and ease of use in secondary analyses.
  Access Control: Access to the shared IPD will be granted to qualified researchers who provide a valid research proposal and agree to comply with data use agreements that ensure the data will be used solely for research purposes and not for commercial gain.
Supporting Information: Study Protocol
Time Frame: Beginning 1 year after publication with no end date.
Access Criteria: Access Control: Access to the shared IPD will be granted to qualified researchers who provide a valid research proposal and agree to comply with data use agreements that ensure the data will be used solely for research purposes and not for commercial gain.

REFERENCES:
- [Background] Lind RR, Geertsen SS, Orntoft C, Madsen M, Larsen MN, Dvorak J, Ritz C, Krustrup P. Improved cognitive performance in preadolescent Danish children after the school-based physical activity programme "FIFA 11 for Health" for Europe - A cluster-randomised controlled trial. Eur J Sport Sci. 2018 Feb;18(1):130-139. doi: 10.1080/17461391.2017.1394369. Epub 2017 Nov 21. PMID 29161988
- [Background] Madsen M, Elbe AM, Madsen EE, Ermidis G, Ryom K, Wikman JM, Rasmussen Lind R, Larsen MN, Krustrup P. The "11 for Health in Denmark" intervention in 10- to 12-year-old Danish girls and boys and its effects on well-being-A large-scale cluster RCT. Scand J Med Sci Sports. 2020 Sep;30(9):1787-1795. doi: 10.1111/sms.13704. Epub 2020 May 27. PMID 32353906